CLINICAL TRIAL: NCT03623893
Title: A Randomized Controlled Trial to Study the Effectiveness and Cost-effectiveness of Contralateral Surgical Exploration During Unilateral Inguinal Hernia Repair in Children.
Brief Title: Hernia Exploration oR Not In Infants Analysis
Acronym: HERNIIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, K.M.A. Dreuning, Coordinating Investigator HERNIIA trial, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017.596; 852001903 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2018-08-02; First posted 2018-08-09 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Inguinal Hernia
Keywords: Metachronous contralateral inguinal hernia; Hernia repair; Contralateral exploration; Cost-effectiveness; Infants
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and care providers are aware of allocation; masking is impossible because of the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Unilateral inguinal hernia repair with contralateral exploration.
  Interventions: Procedure: Contralateral exploration
- Control group (No Intervention): Unilateral inguinal hernia repair.

INTERVENTIONS:
Procedure: Contralateral exploration — Surgery eventually performed when a patent processus vaginalis or hernia exists on the other side than the side on which the child has to be operated on, will be exactly the same as the inguinal hernia repair on the 'symptomatic' side. Exploration of the contralateral side will increase anaesthesia time by 10-15 minutes.
  Arms: Intervention group

SUMMARY:
This study evaluates the effectiveness and cost-effectiveness of contralateral surgical exploration during unilateral inguinal hernia repair in children younger than six months with a unilateral inguinal hernia. In half of the participants contralateral exploration will be performed, while in the other half only unilateral inguinal hernia repair will be performed.

DETAILED DESCRIPTION:
There is a high incidence of metachronous (i.e. a second) contralateral inguinal hernia (MCIH) in infants with an inguinal hernia (5-30%, most studies report 10%), with the highest risk in infants aged less than 6 months. Metachronous hernia is associated with the risk of incarceration and general risks and costs of a second operation. This can potentially be avoided by contralateral exploration at the first operation. On the other hand contralateral exploration may turn out to be unnecessary, is associated with additional operating time and cost, and may be associated with additional complications of surgery (including testicular atrophy, wound infection) and anesthesia. Both policies to routinely explore the contralateral side or not are used in the treatment of unilateral inguinal hernias in children. There is no high-grade level of evidence of the superiority of one of either policy.

ELIGIBILITY:
Inclusion Criteria:

Infants aged younger than six months at first presentation with a primary unilateral inguinal hernia undergoing open hernia repair are considered eligible for inclusion.

Exclusion Criteria:

Infants with (1) incarcerated inguinal hernia requiring urgent surgery, (2) a ventricular-peritoneal drain, (3) non-descended testis.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 416 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Proportion of infants that undergo a second operation | One year after primary hernia repair
  The number of infants that undergo a second operation related to unilateral inguinal hernia within one year after primary inguinal hernia repair

SECONDARY OUTCOMES:
Total duration of operation(s) including anaesthesia time and hospital admission(s) | One year after primary hernia repair
  Total duration of operation(s) including anaesthesia time and total duration of hospital admission(s) related to inguinal hernia within one year after primary repair
Complications of anaesthesia and surgery | During hospital admission, four weeks and one year after primary hernia repair
  Occurence of wound infection, hematoma, hydrocele, testicular atrophy, apnoea or recurrence of inguinal hernia, related to hernia repair.
Health-related quality of life (HRQOL) of the operated infant | At baseline before surgery, 4 weeks and one year after primary hernia repair and, if relevant, four weeks after re-operation
  HRQOL of the operated infants is measured by the TAPQOL (TNO-AZL Preschool Children Quality of Life), a parent-reported questionnaire that is clustered into 12 multi-item scales, with higher scores (range 0-100) indicating better HRQOL.
Parental distress and anxiety | At baseline before surgery, 4 weeks and one year after primary hernia repair and, if relevant, before and four weeks after re-operation
  Parental distress and anxiety of the families of the operated infants is measured by 1) State-Trait Anxiety Inventory (STAI), used as an indicator of parental distress, and 2) Distress Thermometer for Parents (DT-P), a well-validated, brief screening instrument that is frequently used in clinical practice in the Netherlands as a quick screener to identify distress and everyday problems in parents of children who need medical treatment.

OTHER OUTCOMES:
Economic evaluation | Four weeks and one year after primary hernia repair and, if relevant, four weeks after re-operation
  Total health care costs associated with each strategy, assessed by a retrospective cost questionnaire and the iMTA Productivity Cost Questionnaire (iPCQ).

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (7):
  - Amsterdam UMC, Vrije Universiteit Amsterdam, Amsterdam
  - Emma Children's Hospital, Amsterdam UMC, University of Amsterdam, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center, Maastricht
  - Erasmus MC - Sophia Children's Hospital, Rotterdam
  - Juliana Children's Hospital, HagaZiekenhuis, The Hague
  - Máxima Medical Center, Veldhoven

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Dreuning KMA, van Tulder MW, Been JV, Rovers MM, de Graaff JC, Stevens MF, Anema JR, Twisk JWR, van Heurn LWE, Derikx JPM; HERNIIA study group. Contralateral surgical exploration during inguinal hernia repair in infants (HERNIIA trial): study protocol for a multi-centre, randomised controlled trial. Trials. 2021 Sep 30;22(1):670. doi: 10.1186/s13063-021-05606-w. PMID 34593022